CLINICAL TRIAL: NCT04167787
Title: Intelligent Operating Room (InOR) for Orthopaedic Surgery
Acronym: InOR
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Digital Surgery Ltd. (Industry)
Collaborators: University College London Hospitals (Other)
Responsible Party: Sponsor
Other Study IDs: ULCH DS 001
Record Dates: First submitted 2019-10-18; First posted 2019-11-19 (Actual); Last update posted 2019-11-20 (Actual); Status verified 2019-11

CONDITIONS: Knee Replacement; Musculoskeletal
Keywords: Surgery

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The objective of the study is to evaluate the usefulness of digital technologies to support surgical teams before, during, and after an operation.

ELIGIBILITY:
* Inclusion Criteria:
* Adult patients 18-99 years.
* All willing patients undergoing elective total and unicondylar knee replacement (both navigated and robotic-assisted).
* Exclusion Criteria:
* Patients/staff who are unwilling to participate in the study
* Patients/staff that withdraw from the study
* Two stage revisions for infected primary total knee replacements, multiple stage procedures for complex deformities,
* Single stage revision procedures with the need for special instruments and modified steps
* Patients with cognitive impairment/ special cognitive needs.
* <18 years old

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: -Adult patients undergoing elective total and unicondylar knee replacement.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2019-10-10 (Actual); Primary Completion 2020-12-02 (Estimated); Study Completion 2020-12-02 (Estimated)

PRIMARY OUTCOMES:
Change in baseline scores of qualitative questionnaires (every 8 weeks in one surgical team). | 14 months
  To determine how digital technologies and advanced data analytics can improve team coordination, efficiency and performance intraoperatively through understanding and mapping of surgical workflows and instrumentation use.

SECONDARY OUTCOMES:
Report the effect of presenting information intraoperatively through digital displays and augmented reality headsets. | 14 months
  Assessed through monitoring scores from qualitative questionnaires of the surgical team;
To provide automatic post-operative analytics after each surgical operation (up to 150 cases). | 14 months
  Including phase timings and instrumentation

CONTACTS AND LOCATIONS:
Locations (1):
- University College London Hospital NHS Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No